CLINICAL TRIAL: NCT03050294
Title: Study to Evaluate Resistant Disease/Max Adherence to Topical Treatments in Patients With Atopic Dermatitis and Psoriasis
Brief Title: Evaluating Treatment Resistant Dermatitis TaroIIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00039302
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2018-06-15 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis | interventions — Desoximetasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control- Atopic Dermatitis (Active Comparator): Participants with atopic dermatitis will receive desoximetasone and no calls.
  Interventions: Drug: Desoximetasone 0.25% spray
- Atopic Dermatitis Intervention (Experimental): Participants with atopic dermatitis will receive desoximetasone and will be called twice each day, morning and evening, at predetermined times to go over their use of the medication.
  Interventions: Behavioral: Phone calls; Drug: Desoximetasone 0.25% spray
- Control- Psoriasis (Active Comparator): Participants with psoriasis will receive desoximetasone and no calls.
  Interventions: Drug: Desoximetasone 0.25% spray
- Psoriasis Intervention (Experimental): Participants with psoriasis will receive desoximetasone and will be called twice each day, morning and evening, at predetermined times to go over their use of the medication.
  Interventions: Behavioral: Phone calls; Drug: Desoximetasone 0.25% spray

INTERVENTIONS:
Behavioral: Phone calls — Phone calls twice daily
  Arms: Atopic Dermatitis Intervention; Psoriasis Intervention
Drug: Desoximetasone 0.25% spray — Desoximetasone 0.25% spray applied twice daily

SUMMARY:
Psoriasis and atopic dermatitis are chronic inflammatory disease that account for a significant amount of patients in most dermatological practices. Topical corticosteroid agents are often prescribed for treatment of both these conditions, especially when they are localized rather than wide spread. The development of resistance to treatment is termed tachyphylaxis. Poor adherence, rather than down regulation of receptors, may be the primary cause of tachyphylaxis to topical corticosteroids. The primary objective of the study is to determine, under conditions designed to assure good adherence, whether topical 0.25% desoximetasone spray improves clinical outcomes in patients who have resistant inflammatory skin disease defined by failure of previous topical steroid treatment.

DETAILED DESCRIPTION:
Psoriasis and atopic dermatitis are chronic inflammatory disease that account for a significant amount of patients in most dermatological practices. Topical corticosteroid agents are often prescribed for treatment of both these conditions, especially when they are localized rather than wide spread. Prolonged treatment with corticosteroids occasionally results in resistance to treatment. The development of resistance to treatment is termed tachyphylaxis. Tachyphylaxis has been thought to be a result of down regulation of target receptors, resulting is a decreased metabolic effect of the compound.

Poor adherence, rather than down regulation of receptors, may be the primary cause of tachyphylaxis to topical corticosteroids. Patients' use of topical medications decrease over time. Topical spray vehicles have become increasingly more popular because of their rapid application and ease of use. Desoximetasone 0.25% spray is a well-tolerated, FDA approved, potent topical corticosteroid that rapidly and successfully treats inflammatory skin diseases.

Lots of treatment options exist for psoriasis; however, some patients do not get better using these medications. These patients are said to have resistant disease. In this study, we define resistant disease by failure of previous topical steroid treatment. Poor adherence is a barrier to positive clinical outcomes. Failure to respond to medication may be a result of poor adherence rather than resistance to the topical therapy. The purpose of this study is to delineate between the two.

The primary objective of the study is to determine, under conditions designed to assure good adherence, whether topical 0.25% desoximetasone spray improves clinical outcomes in patients who have resistant inflammatory skin disease defined by failure of previous topical steroid treatment.

We propose to enroll 12 subjects with psoriasis and 12 subjects with atopic dermatitis who have "failed" previous topical treatment. Subjects will be required to have body surface area involvement that can be reasonably treated with topical treatment. At the baseline visit, patients will be given Topicort spray and will be shown how to use it. Patients will apply the medication at the initial visit under supervision. Subjects with atopic dermatitis will be treated for 1 week; subjects with psoriasis will be treated for 2 weeks. Visits will take place at baseline, 3 days, 1 week, and in the case of psoriasis, 2 weeks. All subjects enrolled in the study will receive nominal compensation per visit.

To assure good adherence to treatment, patients will be called twice each day, morning and evening, at predetermined times to go over their use of the medication. Disease severity will be measured by EASI (atopic dermatitis)/PASI (psoriasis), Investigator Global Assessment (IGA), and Pruritus Visual Analog Scale (Pruritus VAS). Based on our previous experience, we expect rapid improvement in disease severity measures with good adherence to short term use of highly effective topical treatment. Mean and median changes in the efficacy measures will be reported. In the primary analyses, Wilcoxon signed rank tests will be used to analyze improvements in assessments at end of study compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥18 years of age at baseline visit.

Documentation of plaque-type psoriasis or atopic dermatitis diagnosis as evidenced by one or more clinical features

Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.

Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

No access to a phone throughout the day

Subject is diagnosed with a disease that is known to effect adherence and would otherwise bias our results (Such as Alzheimer's or dementia)

Patient had a history of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance that, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention | Control- Psoriasis | Psoriasis Intervention
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention | Control- Psoriasis | Psoriasis Intervention | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Full Range); unit: years] | 52.8 [27 to 70] | 48 [22 to 67] | 58.3 [40 to 68] | 61.8 [48 to 73] | 55.23 [22 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 3 | 13
  Male | 3 | 3 | 2 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 0 | 7
  White | 2 | 1 | 5 | 6 | 14
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment- Atopic Dermatitis
Description: Investigator's Global Assessment of atopic dermatitis integrates all lesions for overall score. This measure is commonly used to quantify disease severity and most resembles assessments performed in the clinic setting. Score ranges from '0' = Clear to '5' = Very Severe Disease
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 1.7 (0.8) | 1.5 (1.4)

2. Primary Outcome: Investigator Global Assessment- Psoriasis
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Psoriasis | Psoriasis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 2.5 (0.8) | 2.3 (0.5)

3. Secondary Outcome: Total Lesion Severity Score- Atopic Dermatitis
Description: The total lesion severity score measures scaling, erythema, and plaque elevation. The score range is 0-15, with higher scores denoting worse outcomes.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 3.8 (2.5) | 4.7 (5.6)

4. Secondary Outcome: Total Lesion Severity Score-Psoriasis
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Psoriasis | Psoriasis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 6.5 (3.1) | 5.8 (1.3)

5. Secondary Outcome: Eczema Area and Severity Index- Atopic Dermatitis
Description: Eczema Area and Severity Index (EASI): Disease severity will be assessed by a physician with the Eczema Area and Severity Index (EASI). This measure is commonly used and well validated instrument of eczema severity. It is weighted for area in each of the four body regions (which differs for adults and children under 7) and scores erythema, excoriation, induration/papulation, and lichenification. The total scores range from 0-72. Higher scores represent more severe eczema.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 3.1 (5.1) | 1.2 (1.1)

6. Secondary Outcome: Pruritus Visual Analog Scale- Atopic Dermatitis
Description: The Pruritus VAS is a scale consisting of a 10cm long line and a single question. The left end point represents "no itch" (score of 0) and the right end point the "worst imaginable itch" (score of 10).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 1.1 (2.0) | 1.2 (1.2)

7. Secondary Outcome: Pruritus Visual Analog Scale- Psoriasis
Description: as for outcome 6
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Psoriasis | Psoriasis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 1.4 (0.9) | 1.3 (1.3)

8. Secondary Outcome: Psoriasis Area and Severity Index
Description: The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected areas (head, arms, trunk, and legs). The severity of three clinical signs (erythema, induration and desquamation) are on a scale from 0 to 4 (from absent to very severe). An area and severity score for each region is calculated by multiplying the area score by the severity score. The score range is 0-72, with higher scores denoting worse outcomes.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control- Psoriasis | Psoriasis Intervention
Number analyzed (Participants) | 6 | 6
units on a scale | 7.1 (5.1) | 5.1 (3.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Control- Atopic Dermatitis | Atopic Dermatitis Intervention | Control- Psoriasis | Psoriasis Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03050294/Prot_SAP_000.pdf